CLINICAL TRIAL: NCT06931431
Title: UNCPM 22322 - Adaption of the Transition of Care Model for Post-Discharge HIV-NCD Care in Lilongwe, Malawi - MLATHO
Acronym: MLATHO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-2753; 1R21TW012647-01 (NIH)
Record Dates: First submitted 2025-04-14; First posted 2025-04-17 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: HIV; Noncommunicable Diseases
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: The Transition of Care Model (TCM) is an evidence-based model in the United States of America (USA) focused on continuity of care for patients with complex needs, particularly mature adults, as they move through the health care system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transition of Care Model (TCM) (Experimental): Following hospitalization for comorbid HIV and non-communicable diseases, participants will be followed for 3 months post discharge using the adopted Transition of Care Model (TCM).
  Interventions: Behavioral: Transition of Care Model (TCM)

INTERVENTIONS:
Behavioral: Transition of Care Model (TCM) — Key components of the TCM include discharge assessment, care planning, provider communication with outpatient follow-up teams, and community-based follow-up

SUMMARY:
This is an implementation research study that will adapt and pilot test the Transitional Of Care Model (TCM), originally conceived and developed in the USA, for targeted use as a post-discharge intervention for adults hospitalized with comorbid HIV and NCDs in Malawi using a mixed methods approach.

DETAILED DESCRIPTION:
This study will enroll 75 consecutive adults hospitalized with comorbid HIV and at least have one common cardiometabolic condition (e.g., hypertensive urgency, heart failure, stroke, or diabetes) and provide them with the adapted TCM according to the SOP developed in the prior phase. It is expected that 15-20% will also have comorbid opportunistic infections.

The study will evaluate the acceptability and feasibility of the adapted intervention.

Using mixed methods, including surveys and interviews, the study will evaluate the acceptability and feasibility of providing the inpatient and post-discharge components of the adapted TCM. The study will also describe key 3-month post-discharge clinical outcomes (mortality, readmission) and indicators that may mediate clinical outcomes (linkages/retention in care, adherence to antiretroviral therapy/non-communicable disease (ART/ NCDs) medications, dual control of HIV and NCDs, social demographic variables). Clinical outcomes and indicators in the pilot participants will be compared with a comparable historical control group of patients who had routine care at KCH in the recent past.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* living with HIV
* admitted to internal medicine
* has at least a cardiometabolic NCO as the primary or secondary reason for admission based on the HIV inpatient consultation

Exclusion Criteria:

* patients living beyond Lilongwe urban

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Post-discharge home visits | Through 3-months post-discharge
  Proportion of discharged participants who have a home visit by a nurse within 1 week of discharge
Completion of comprehensive needs assessment | Through 3-months post-discharge
  Proportion of participants who have an assessment of social support, food insecurity, medication adherence self-efficacy during hospitalization or within 1 week of discharge
Feasibility rating from health worker perspective. | At 3 months post-discharge
  Feasibility of intervention measure (FIM) score among health workers involved in the implementation of the post-discharge intervention.The FIM is a 4-item/ statement measure
  1. The post-discharge intervention program seems implementable in our setting
  2. The post-discharge intervention seems possible in our setting
  3. The post-discharge intervention seems doable in our setting
  4. The post-discharge intervention seems easy to use for our setting The FIM is measured on a five-point rating scale:( 1= completely disagree, 2= disagree,3=neither agree nor disagree, 4= agree, and 5 = completely agree) The mean score ranges from 1 to 5, with 1 indicating the least feasibility and 5 indicating the most feasibility.
Feasibility rating from patient and caregiver perspective | At 3 months post-discharge
  Feasibility of implementation measure (FIM) score among patients and caregivers who were assigned to receive the post-discharge intervention.The FIM is a 4-item/ statement measure
  1. The post-discharge intervention program seems implementable in our setting
  2. The post-discharge intervention seems possible in our setting
  3. The post-discharge intervention seems doable in our setting
  4. The post-discharge intervention seems easy to use for our setting The FIM is measured on a five-point rating scale:( 1= completely disagree, 2= disagree,3=neither agree nor disagree, 4= agree, and 5 = completely agree) The mean score ranges from 1 to 5, with 1 indicating the least feasibility and 5 the most feasibility.
Reach among eligible hospitalized adults with HIV/NCD comorbidity | At completion of enrollment
  Proportion of eligible adults admitted with HIV/NCD comorbidity who participate in the study during the enrollment period
Acceptability of Intervention Measures(AIM) rating from patient and caregiver perspective | At 3 months post-discharge
  The AIM is a 4-item/ statement measure
  1. The post-discharge intervention implementation program meets my approval
  2. The post-discharge intervention is appealing to me
  3. I like the post-discharge intervention
  4. I welcome the post-discharge intervention The AIM is measured on a five-point rating scale:( 1= completely disagree, 2= disagree,3=neither agree nor disagree, 4= agree, and 5 = completely agree) The mean score ranges from 1 to 5, with 1 indicating poorly acceptable and five highly acceptable
Acceptability of Intervention Measures(AIM) rating from Healthcare Workers perspective | At 3 months post-discharge
  The AIM is a 4-item/ statement measure
  1. The post-discharge intervention implementation program meets my approval
  2. The post-discharge intervention is appealing to me
  3. I like the post-discharge intervention
  4. I welcome the post-discharge intervention The AIM is measured on a five-point rating scale:( 1= completely disagree, 2= disagree,3=neither agree nor disagree, 4= agree, and 5 = completely agree) The mean score ranges from 1 to 5, with 1 indicating poorly acceptable and 5 highly acceptable.
Intervention Appropriateness Measure(IAM) rating from Healthcare Workers perspective | At 3 months post-discharge
  The IAM is a 4-item/ statement measure
  1. The post-discharge intervention program seems fitting in our setting
  2. The post-discharge intervention seems suitable for our setting
  3. The post-discharge intervention seems applicable to our setting
  4. The post-discharge intervention seems a good match in our setting The IAM is measured on a five-point rating scale:( 1= completely disagree, 2= disagree,3=neither agree nor disagree, 4= agree, and 5 = completely agree) The mean score ranges from 1 to 5, with 1 indicating the least appropriate and 5 the most appropriate
Intervention Appropriateness Measure(IAM) rating for patient and caregiver | At 3 months post-discharge
  The IAM is a 4-item/ statement measure
  1. The post-discharge intervention program seems fitting in our setting
  2. The post-discharge intervention seems suitable for our setting
  3. The post-discharge intervention seems applicable to our setting
  4. The post-discharge intervention seems a good match in our setting The IAM is measured on a five-point rating scale:( 1= completely disagree, 2= disagree,3=neither agree nor disagree, 4= agree, and 5 = completely agree) The mean score ranges from 1 to 5, with 1 indicating the least appropriate and 5 the most appropriate.

SECONDARY OUTCOMES:
The number of participants re-hospitalization after discharge | Through 3 months post-discharge
  Proportion of participants who are discharged and then readmitted
Dual control of HIV and hypertension | At 3 months post-discharge
  Among participants with hypertension and HIV, the proportion with both HIV viral load below assay detection (<40 copies/ml) and blood pressure below 140/90
Dual control of HIV and diabetes | At 3 months post-discharge
  Among participants with diabetes and HIV, the proportion with HIV viral load below assay detection (<40 copies/ml) and hemoglobin A1C <7%
Control of hypertension | At 3 months post-discharge
  Among participants with hypertension, the proportion with blood pressure below 140/90
Control of diabetes | At 3 months post-discharge
  Among participants with diabetes, the proportion with hemoglobin A1C <7%
HIV viral suppression | At 3 months post-discharge
  The proportion with HIV viral load below assay detection (<40 copies/ml)
All-cause post-discharge mortality | Through 3-months post-discharge
  The proportion with death after discharge from the index admission

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Kanyama, MBBS, Principal Investigator — University of North Carolina at Chapel Hill (Project Malawi)
Locations (1):
- Kamuzu Central Hospital, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
  More information provided by University of North Carolina, Chapel Hill
Supporting Information: Study Protocol
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.
URL: http://unc.edu